CLINICAL TRIAL: NCT00816205
Title: An Open Label Study to Examine the Effect of Coated Nifedipine Suppositories on Anal Pressure in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Michael Shapiro MD, Gastroenterology Dept, Asaf Harofe Medical Center
Allocation: Not Applicable | Model: Single Group
Other Study IDs: RDD102
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Anal Resting Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): This is an open label, dose-finding study. After detrminig baseline resting anal pressure with a manometric test, coated Suppositories will be administered intra rectally. Subjects will take rectally a total of 3 Coated Suppositories per study.
  Interventions: Drug: Coated Nifedipine Suppositories

INTERVENTIONS:
Drug: Coated Nifedipine Suppositories — Subjects will take rectally a total of 3 Coated Suppositories per study. 90 minutes after each coated suppository insertion this suppository will be removed and a amnometric study will be performed:
  The first dose will contain 4 mg of Nifedipine and the manomentric measurement performed afterwards will be used to determine baseline anal pressures.
  The second dose will contain 12 mg of Nifedipine. The third dose will contain 24 mg of Nifedipine.

SUMMARY:
This is an open label, dose-finding study. Approximately 8 healthy subjects will be participating in this study.

Within one week after the screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will enter a one day treatment period. During this period, 4 anal manometric studies will take place. Study medication (Coated Nifedipine suppositories at various doses) will be administered at pre-determined intervals. During the study, blood samples will be obtained for plasma Nifedipine analysis.

DETAILED DESCRIPTION:
After detrminig baseline resting anal pressure with a manometric test, coated Suppositories will be administered intra rectally. Subjects will take rectally a total of 3 Coated Suppositories per study. 90 minutes after each coated suppository insertion this suppository will be removed and a amnometric study will be performed:

The first dose will contain 4 mg of Nifedipine and the manomentric measurement performed afterwards will be used to determine baseline anal pressures.

The second dose will contain 12 mg of Nifedipine. The third dose will contain 24 mg of Nifedipine. The primary efficacy parameter is change in Resting Anal Pressure from baseline.

The secondary efficacy parameters include the following:

* The ratio of change in anal pressure to plasma Nifedipine level.
* The ratio of change in anal pressure to change in blood pressure.
* The ratio of change in anal pressure to change in heart rate.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria will be eligible to participate in the trial:

* Signed written informed consent;
* Male or female subjects 18 to 55 years of age;

Exclusion Criteria:

Subjects are excluded from participation in the study if any of the following criteria apply:

Has a clinically significant history or presence of any of the following conditions:

* Known allergy to Nifedipine, polyethylene-glycol, Propylene-glycol or silicone.
* Active or past history of disease that requires medication or clinical follow up.
* Malignant disease within 5 years of screening;
* History of ano rectal disease.
* History of gastrointestinal disease.
* History of gastrointestinal bleeding.
* History of rectal surgery.
* History of gastrointestinal surgery.
* History of HIV.
* In need of chronic use of medication, with the exception of birth control medications.
* Currently uses medication for acute illness.
* Has upon physical examination a rectal deformation or signs of rectal disease such as fissure, bleeding hemorrhoids, fistula., infection or space occupying lesion.
* Has received any investigational drug within 90 days of screening;
* Receipt of any investigational treatment (drug or device) within 90 days prior to screening;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is change in Resting Anal Pressure from baseline. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Gastroeneterology, Asaf Harofe Medical Center, Zrifin, Israel